CLINICAL TRIAL: NCT01523821
Title: Treatment of Steroid Non-responsive Acute GVHD With Alpha 1 Antitrypsin (AAT). A Phase I/II Study
Brief Title: Alpha 1 Anti-Trypsin (AAT) in Treating Patients With Acute Graft-Versus-Host Disease GVHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2571.00; NCI-2011-03805 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2571; 2571.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01HL036444 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2012-01-23; First posted 2012-02-01 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Graft-Versus-Host Disease (GVHD) Acute on Chronic
MeSH Terms: conditions — Graft vs Host Disease | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Intervention Model Description: The study will have three escalating alpha 1 anti-trypsin (AAT) dose cohorts with six patients in each cohort (Phase I). Based on response and toxicity, an additional six patients will be enrolled in the optimal dose (Phase II).
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (30 mg/kg) (Other): Alpha 1 anti-trypsin (AAT) will be administered intravenously at a dose of 90 mg/kg (loading dose) on day 1 followed by 30mg/kg (maintenance dose) every other day (QOD) on days 3, 5, 7, 9, 11, 13 & 15.
  Interventions: Drug: Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia]
- Cohort 2 (60 mg/kg) (Other): AAT will be administered intravenously at a dose of 90 mg/kg (loading dose) on day 1 followed by 60 mg/kg (maintenance dose) QOD on days 3, 5, 7, 9, 11, 13 & 15.
  Interventions: Drug: Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia]
- Cohort 3 (90 mg/kg) (Other): AAT will be administered intravenously at a dose of 90 mg/kg on days 1, 3, 5, 7, 9, 11, 13 & 15.
  Interventions: Drug: Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia]

INTERVENTIONS:
Drug: Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia] — Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia] at various levels over different days

SUMMARY:
This phase I/II trial evaluates the efficacy and adverse effects of alpha 1 anti-trypsin (AAT) for the treatment of acute graft-versus-host disease (GVHD) after hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of AAT in patients with steroid non-responsive acute GVHD.

II. Characterize pharmacodynamic effects of AAT on pro-inflammatory cytokines, heparan sulfate, and the spectrum of peripheral blood T cells.

III. Determine clinical responses of GVHD to AAT in patients with steroid non-responsive acute GVHD.

OUTLINE: This is a phase I/II dose-escalation study of AAT.

Patients will receive AAT intravenously (IV) on study days 1, 3, 5, and 7. Patients who experience no toxicity and in whom GVHD is stable or improved after the day 7 dose can continue therapy with AAT on days 9, 11, 13 and 15 for a total of 8 doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted from related or unrelated, human leukocyte antigen (HLA) matched or mismatched donors
* Patients transplanted with hematopoietic stem cells from any source
* Patients receiving calcineurin inhibitors as part of graft versus host disease (GVHD) prophylaxis
* Patients with acute GVHD grades II-IV developing despite GVHD prophylaxis
* Patients who have not shown a satisfactory response to methylprednisolone-equivalent doses at 2 mg/kg/day, based on adjusted body weight
* Signed and dated informed consent

Exclusion Criteria:

* Patients who have received any systemic agents in addition to steroids for treatment of GVHD
* Patients unable to give informed consent
* Patients with manifestations of classic chronic GVHD
* Patients with evidence of recurrent malignancy
* Patients with acute/chronic GVHD overlap syndrome
* Patients whose GVHD developed after donor lymphocyte infusion (DLI)
* Patients with severe organ dysfunction, defined as

  * On dialysis
  * Requiring oxygen (O2) at more than 2 l/min
  * Uncontrolled arrhythmia or heart failure
  * Veno-occlusive disease (sinusoidal obstruction syndrome)
* Patients with uncontrolled infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10-11 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Joachim Deeg, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients signed IRB-approved consents during the period of 12/11/13 to 12/22/16. Treatment with alpha 1 anti-trypsin (AAT) typically started within 24 hours of consent. Patients were identified by clinical staff as needing additional treatment for acute graft versus his disease (GVHD) following initial therapy with corticosteroids.
Groups:
- Cohort 1 (30 mg/kg): AAT will administered intravenously at a dose of 90 mg/kg (loading dose) on day 1 followed by 30mg/kg (maintenance dose) QOD on days 3, 5, 7, 9, 11, 13 & 15.
  Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia]
- Cohort 2 (60 mg/kg): AAT will be administered intravenously at a dose of 90 mg/kg (loading dose) on day 1 followed by 60 mg/kg (maintenance dose) QOD on days 3, 5, 7, 9, 11, 13 & 15.
  Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia]
- Cohort 3 (90 mg/kg): AAT will be administered intravenously at a dose of 90 mg/kg on days 1, 3, 5, 7, 9, 11, 13 & 15.
  Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia]
Period: Overall Study
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg)
Started | 8 | 6 | 6
Completed | 8 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 (30 mg/kg): AAT will be administered intravenously at a dose of 90 mg/kg (loading dose) on day 1 followed by 30mg/kg (maintenance dose) QOD on days 3, 5, 7, 9, 11, 13 & 15.
  Alpha 1-Proteinase Inhibitor, Human 1 MG [Glassia]
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg) | Total
Number analyzed (Participants) | 8 | 6 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 6 | 18
  >=65 years | 0 | 2 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 49 [23 to 59] | 40 [26 to 73] | 51 [38 to 63] | 48 [23 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 6 | 9
  Male | 5 | 6 | 0 | 11
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number (Percentage) of Patients at Each Dosing Cohort Who Experience no Toxicity and in Whom Graft Versus Host Disease (GVHD) is Stable or Improved
Description: Toxicity and adverse events were assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. All adverse events were reported regardless of attribution to alpha 1 anti-trypsin (AAT). GVHD response was defined per standard criteria for improvement, no change or progression of signs/symptoms in skin rash (% body surface area), GI (nausea, vomiting, anorexia, diarrhea, GI bleeding, abdominal cramping) and hepatic function (serum bilirubin levels). For this outcome measure, the requirement for additional GVHD treatment beyond AAT was not included in the criteria for response (i.e patients who may have required additional GVHD treatment before study day 28 were not automatically categorized as non-responders or as having progressive GVHD).
Time Frame: Adverse events were reported through 15 days after the last dose of AAT. GVHD response assessed at study day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg)
Number analyzed (Participants) | 8 | 6 | 6
Participants | 6 | 2 | 2

2. Secondary Outcome: Number (Percentage) of Patients at Each Dosing Cohort Experiencing an Unexpected Serious Adverse Event (SAE)
Description: Serious adverse events included death, a life-threatening adverse drug experience, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/ incapacity, or congenital anomaly/birth defect. Significant events that do not meet these criteria may be considered serious if they jeopardize the patient and require a medical intervention to prevent one of the outcomes above. An "unexpected" adverse event is defined as an event that is not identified in nature, severity or frequency in the current investigator brochure/package insert/product information.
Time Frame: SAEs were reported through 30 days after the last dose of alpha 1 anti-trypsin (AAT).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg)
Number analyzed (Participants) | 8 | 6 | 6
Participants | 2 | 0 | 0

3. Secondary Outcome: Number (Percentage) of Patients at Each Dosing Cohort Who Experience One or More Suspected Serious Adverse Reactions (Infusion Related Reactions)
Description: Serious adverse reactions were assessed by the NCI CTCAE v4.0.
Time Frame: Within 48 hours after each infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg)
Number analyzed (Participants) | 8 | 6 | 6
Participants | 0 | 0 | 0

4. Secondary Outcome: Number (Percentage) of Patients at Each Dosing Cohort Who Experience One or More Thrombotic or Thrombo-embolic Events
Description: Events were assessed using the NCI CTCAE v4.0.
Time Frame: Events were reported through 15 days after the last dose of AAT.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg)
Number analyzed (Participants) | 8 | 6 | 6
Participants | 0 | 0 | 0

5. Secondary Outcome: Number (Percentage) of Patients at Each Dosing Cohort With Occurrence of Infections
Description: Infections were assessed using NCI CTCAE v4.0.
Time Frame: Infections were reported through 15 days after the last dose of AAT.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg)
Number analyzed (Participants) | 8 | 6 | 6
Participants | 7 | 5 | 5

6. Secondary Outcome: Number (Percentage) of Patients at Each Dosing Cohort With Progression of GVHD
Description: GVHD responses were assessed using criteria established by the Center for International Blood and Marrow Transplant Research and criteria from the Acute GVHD Activity Index. Patients who required additional systemic GVHD treatment beyond AAT before study day 28 were defined as having progressive GVHD.
Time Frame: GVHD responses were assessed on day 28 after starting AAT therapy or at time of death if patient died before study day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg)
Number analyzed (Participants) | 8 | 6 | 6
Participants | 4 | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were reported through 15 days after the last dose of AAT. Serious adverse events were reported if they occurred within 30 days after the last dose of AAT.
Description: All adverse events were collected regardless of attribution to AAT. Included are events that worsened from baseline.
Arm/Group | Cohort 1 (30 mg/kg) | Cohort 2 (60 mg/kg) | Cohort 3 (90 mg/kg)
All-Cause Mortality (participants affected / at risk) | 6/8 | 4/6 | 4/6
Serious Adverse Events (participants affected / at risk) | 8/8 | 5/6 | 4/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (30 mg/kg) (N=8) | Cohort 2 (60 mg/kg) (N=6) | Cohort 3 (90 mg/kg) (N=6)
acute graft-versus-host disease (Immune system disorders) | 2 | 4 | 3
infection (Infections and infestations) | 1 | 1 | 1
perirectal abbess (Gastrointestinal disorders) | 1 | 0 | 0
bowel perforation (Gastrointestinal disorders) | 1 | 0 | 0
liver failure (Hepatobiliary disorders) | 1 | 0 | 0
diffuse alveolar hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
cranial hemorrhage (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort 1 (30 mg/kg) (N=8) | Cohort 2 (60 mg/kg) (N=6) | Cohort 3 (90 mg/kg) (N=6)
thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6 | 4
hypogammaglobulinemia (Blood and lymphatic system disorders) | 2 | 2 | 2
neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 3
anemia (Blood and lymphatic system disorders) | 2 | 5 | 1
leukocytosis (Blood and lymphatic system disorders) | 2 | 2 | 1
HUS/microangiopathy (Blood and lymphatic system disorders) | 2 | 1 | 2
hyperglycemia (Metabolism and nutrition disorders) | 3 | 2 | 3
hypokalemia (Metabolism and nutrition disorders) | 5 | 2 | 1
hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 0
hypomagnesemia (Metabolism and nutrition disorders) | 6 | 1 | 3
hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 0
elevated LDH (Metabolism and nutrition disorders) | 1 | 0 | 0
hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 2
hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 3
hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
weakness (Musculoskeletal and connective tissue disorders) | 6 | 5 | 5
joint pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
fall (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
edema/fluid overload (Cardiac disorders) | 5 | 5 | 5
hypotension (Cardiac disorders) | 1 | 2 | 2
orthostatic hypotension (Cardiac disorders) | 1 | 3 | 1
bradycardia (Cardiac disorders) | 1 | 0 | 1
hypertension (Cardiac disorders) | 2 | 3 | 0
tachycardia (Cardiac disorders) | 1 | 1 | 2
dehydration (Cardiac disorders) | 0 | 1 | 0
atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
gall bladder sludge (Hepatobiliary disorders) | 1 | 0 | 0
elevated liver function tests (Hepatobiliary disorders) | 2 | 4 | 0
iron overload (Hepatobiliary disorders) | 1 | 0 | 0
ascites (Hepatobiliary disorders) | 0 | 1 | 0
dizziness (Nervous system disorders) | 2 | 1 | 0
neuropathy (Nervous system disorders) | 2 | 0 | 0
tremor (Nervous system disorders) | 2 | 1 | 0
altered mental status (Nervous system disorders) | 1 | 2 | 1
seizure (Nervous system disorders) | 1 | 1 | 0
headache (Nervous system disorders) | 2 | 1 | 1
somnolence (Nervous system disorders) | 0 | 1 | 1
numbness (leg) (Nervous system disorders) | 0 | 0 | 1
blister/excoriation (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
rash/erythema (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
wound (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
pain (all sites combined) (General disorders) | 4 | 2 | 2
anxiety/stress (Psychiatric disorders) | 4 | 1 | 0
depression (Psychiatric disorders) | 3 | 1 | 2
delirium (Psychiatric disorders) | 1 | 0 | 0
lethargy (Psychiatric disorders) | 1 | 0 | 0
gastroesophageal reflux (Gastrointestinal disorders) | 1 | 1 | 1
constipation (Gastrointestinal disorders) | 2 | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
nausea (Gastrointestinal disorders) | 2 | 0 | 0
hemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0
peri-rectal abcess (Gastrointestinal disorders) | 1 | 0 | 0
gastroparesis (Gastrointestinal disorders) | 0 | 2 | 0
peri-rectal irritation (Gastrointestinal disorders) | 0 | 0 | 1
hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
consolidation (on CXR) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
dry mouth (Gastrointestinal disorders) | 1 | 3 | 2
oral lesion/ulcer (Gastrointestinal disorders) | 2 | 0 | 0
oral plaques (Gastrointestinal disorders) | 0 | 1 | 0
dry eyes (Eye disorders) | 1 | 0 | 1
blurred vision (Eye disorders) | 1 | 1 | 0
scleral discharge (Eye disorders) | 1 | 0 | 0
corneal abrasion (Eye disorders) | 0 | 1 | 0
hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1
facial/neck swelling (General disorders) | 1 | 1 | 0
fatigue (General disorders) | 4 | 5 | 4
chills (General disorders) | 1 | 0 | 0
insomnia (General disorders) | 1 | 4 | 1
hiccups (General disorders) | 2 | 1 | 0
dysuria (Renal and urinary disorders) | 2 | 1 | 1
penile lesion (Skin and subcutaneous tissue disorders) | 1/5 | 1 | 0/0
scrotal edema (Renal and urinary disorders) | 1/5 | 2 | 0/0
hematuria (Renal and urinary disorders) | 0 | 2 | 0
acute kidney injury (Renal and urinary disorders) | 3 | 2 | 0
acute graft versus host disease (GVHD) (Immune system disorders) | 2 | 4 | 3
liver failure (Hepatobiliary disorders) | 1 | 0 | 0
bowel perforation (Gastrointestinal disorders) | 1 | 0 | 0
diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
cranial hemorrhage (Nervous system disorders) | 1 | 0 | 0
infection (Infections and infestations) | 7 | 5 | 5
acute myelogenous leukemia (Blood and lymphatic system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No